CLINICAL TRIAL: NCT03800472
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Including the Effect of Food, and Pharmacodynamics of Single and Multiple Ascending Oral Doses of GLPG3312, in Adult, Healthy Subjects
Brief Title: A Study Investigating the Safety, Absorption and Elimination of GLPG3312, a New Drug in the Treatment of Inflammatory Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG3312-CL-101; 2018-001955-11 (EudraCT Number)
Record Dates: First submitted 2019-01-03; First posted 2019-01-11 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part 1 (SAD IR), Part 2 (SAD MR) and Part 4 (MAD MR) are randomized, double-blind, placebo-controlled; Part 3 (FE MR) is open-label.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- GLPG3312 SAD IR (Part 1) (Experimental): Single doses of GLPG3312 IR
  Interventions: Drug: GLPG3312 IR
- Placebo SAD IR (Part 1) (Placebo Comparator): Single doses of Placebo IR
  Interventions: Drug: Placebo
- GLPG3312 SAD MR (Part 2) (Experimental): Single doses of GLPG3312 MR
  Interventions: Drug: GLPG3312 MR
- Placebo SAD MR (Part 2) (Placebo Comparator): Single doses of Placebo MR
  Interventions: Drug: Placebo
- GLPG3312 FE MR (Part 3) (Experimental): Single dose of GLPG3312 MR in fed and fasted state
  Interventions: Drug: GLPG3312 FE MR
- GLPG3312 MAD MR (Part 4) (Experimental): Multiple doses of GLPG3312 MR
  Interventions: Drug: GLPG3312 MR
- Placebo MAD MR (Part 4) (Placebo Comparator): Multiple doses of Placebo MR
  Interventions: Drug: Placebo
- GLPG3312 MAD MR optimized (Part 4) (Experimental): Multiple doses of GLPG3312 MR
  Interventions: Drug: GLPG3312 MR
- Placebo MAD MR optimized (Part 4) (Placebo Comparator): Multiple doses of Placebo MR
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG3312 IR — GLPG3312 IR tablets, up to 4 single ascending oral doses (A, B, C, D).
  Arms: GLPG3312 SAD IR (Part 1)
Drug: Placebo — Placebo tablets
  Arms: Placebo MAD MR (Part 4); Placebo SAD IR (Part 1); Placebo SAD MR (Part 2)
Drug: GLPG3312 MR — GLPG3312 MR film-coated tablets, up to 4 single ascending oral doses (H, I, J, K).
  Arms: GLPG3312 SAD MR (Part 2)
Drug: GLPG3312 FE MR — GLPG3312 MR film-coated tablets, single oral dose (N) on 2 occasions, i.e. in fed state after a high-fat high-calorie breakfast, and in fasted state.
  Arms: GLPG3312 FE MR (Part 3)
Drug: GLPG3312 MR — GLPG3312 MR film-coated tablets, up to 2 multiple ascending oral doses (O, P).
  Arms: GLPG3312 MAD MR (Part 4)
Drug: GLPG3312 MR — GLPG3312 MR optimized film-coated tablets, up to 3 multiple ascending oral doses (Q, R, S).
  Arms: GLPG3312 MAD MR optimized (Part 4)
Drug: Placebo — Placebo optimized tablets
  Arms: Placebo MAD MR optimized (Part 4)

SUMMARY:
The purpose of this study is to investigate how safe 2 different formulations (immediate-release (IR) and modified-release (MR) tablets) of the new compound GLPG3312 are and how well they are tolerated when they are administered to healthy volunteers. Immediate-release and modified-release tablets contain the same active ingredient, but the modified-release tablet is covered with a protective layer, so it will dissolve in the intestines and not in the stomach. GLPG3312 has not been administered to humans before. Next to assessing the safety and tolerability, the purpose of this study is to investigate how food affects how quickly and to what extent GLPG3312 in a modified release formulation is absorbed and eliminated from the body. In addition, the effect of GLPG3312 on the body will be investigated by evaluating the effect of GLPG3312 on markers of the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 to 55 years of age (extremes included), on the date of signing the Informed Consent Form (ICF). Female should be of non-childbearing potential defined as permanently surgically sterile (bilateral oophorectomy, i.e. surgical removal of ovaries, bilateral salpingectomy or hysterectomy, i.e. surgical removal of uterus), or with no menses for 12 or more months without an alternative medical cause AND a folliclestimulating hormone (FSH) level >35 IU/L. These subjects must also have a negative pregnancy test. For surgical sterilization, documented confirmation will be requested.
* A body mass index (BMI) between 18 to 30 kg/m2, inclusive.
* Subject must be able and willing to comply with restrictions on prior medication.
* Male subjects with female partners of childbearing potential must be willing to comply with contraceptive methods.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and fasting clinical laboratory safety tests. Clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered nonclinically significant in the opinion of the investigator. At minimum hemoglobin, alanine aminotransferase (ALT), creatinine, creatine kinase-myoglobin (CK-MB), High Sensitivity Troponin I, Troponin T and alkaline phosphatase must be within the normal range, aspartate aminotransferase (AST) must be no greater than 1.5x upper limit of normal range (ULN).

Exclusion Criteria:

* Known hypersensitivity to IMP ingredients or history of a significant allergic reaction to IMP ingredients as determined by the investigator.
* Positive serology for HBsAg, or hepatitis C virus (HCV), or history of hepatitis from any cause with the exception of hepatitis A that was resolved at least 3 months prior to first dosing of the IMP.
* History of, or a current immunosuppressive condition (e.g. HIV infection).
* Having any illness (e.g. active allergy, fever, hypersensitivity reactions) judged by the investigator as clinically significant, in the 3 months prior to first dosing of the IMP.
* Any history, or current sign or symptom of a cardiovascular, renal, or metabolic bone disease or disease of bone remodelling (with the exception of uncomplicated accidental bone fractures that recovered uncompromised at least 1 year ago), or any history of endocrine disease, including an abnormal laboratory result for prespecified clinical laboratory safety parameters related to these conditions.
* Presence or sequelae of gastrointestinal, liver, kidney (creatinine clearance ≤80 mL/min/1.73m2, using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula: if calculated result is ≤80 mL/min/1.73m2, a 24-hours urine collection can be done), or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of malignancy within the past 5 years prior to screening with the exception of excised and curatively treated non-metastatic cell carcinoma of the skin or carcinoma in situ of the cervix which is considered cured with minimal risk of recurrence.
* Significant blood loss (including blood donation >450 mL), or transfusion of any blood product within 12 weeks prior to screening.
* Treatment with any medication (including over-the-counter and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements) except occasional paracetamol (maximum dose of 2 g/day and a maximum of 10 g/ 2 weeks) in the last 2 weeks or 5 half-lives of the drug, whichever is longer, prior to the first dosing of the IMP.
* Active drug abuse or alcohol abuse (alcohol abuse defined as regular weekly intake of more than 14 units) within 2 years prior to first IMP administration.
* Active smoker and/or has used nicotine or nicotine-containing products within the past 6 months before the first IMP administration.
* Regular consumption of a large quantity of caffeinated coffee, tea (> 6 cups per day) or equivalent.
* Concurrent participation or participation in a drug, drug/device or biologic investigational research study within 12 weeks or 5 half-lives of the IMP, whichever is longer, prior to first dosing of the investigational medicinal product (IMP).
* Any clinical laboratory test result outside of the reference ranges considered by the investigator as clinically significant. Hemoglobin, ALT, creatinine, CK-MB, High Sensitivity Troponin I, Troponin T, or alkaline phosphatase outside normal range, AST result greater than 1.5x ULN.
* History or presence of clinically significant abnormalities detected on 12-lead ECG of either rhythm or conduction (e.g. known long QT syndrome). A first-degree atrioventricular block will not be considered as a significant abnormality. QTcF = QT x (1000/RR)1/3 (QTcF) >450 ms (male), >460 ms (female) (mean values per parameter will be considered) detected on the 12-lead ECG.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment emergent adverse events (TEAEs), treatment-emergent serious adverse events, and TEAEs leading to treatment discontinuations | From screening through study completion, an average of 9 months.
  To evaluate the safety and tolerability of oral single and multiple ascending doses of GLPG3312, in adult, healthy, subjects, when given as Immediate Release (IR) formulation (in fasted conditions) or as Modified Release (MR) formulation (in fasted and fed conditions)

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG3312 (μg/mL) (Part 1) | Between Day 1 pre-dose and Day 4
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3312, in adult, healthy subjects, when given as IR formulation
Maximum observed plasma concentration (Cmax) of GLPG3312 (μg/mL) (Part 2) | Between Day 1 pre-dose and Day 7
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3312, in adult, healthy, subjects, when given as MR formulation
Maximum observed plasma concentration (Cmax) of GLPG3312 (μg/mL) under fed conditions (high-fat high calorie) versus fasted conditions (Part 3) | Between Day 1 pre-dose and Day 7
  To evaluate the food effect on the PK of a single oral dose of GLPG3312 in adult, healthy, subjects, when given as MR formulation
Maximum observed plasma concentration (Cmax) of GLPG3312 (μg/mL) (Part 4) | Between Day 1 pre-dose and Day 21
  To evaluate the pharmacokinetics (PK) of oral MAD of GLPG3312, in adult, healthy, subjects, when given as MR formulation
Area under curve (AUC) of GLPG3312 (μg.h/mL) (Part 1) | Between Day 1 pre-dose and Day 4
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3312, in adult, healthy, subjects, when given as IR formulation
Area under curve (AUC) of GLPG3312 (μg.h/mL) (Part 2) | Between Day 1 pre-dose and Day 7
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3312, in adult, healthy, subjects, when given as MR formulation
Area under curve (AUC) of GLPG3312 (μg.h/mL) under fed conditions (high-fat high calorie) versus fasted conditions (Part 3) | Between Day 1 pre-dose and Day 7
  To evaluate the food effect on the PK of a single oral dose of GLPG3312 in adult, healthy, subjects, when given as MR formulation
Area under curve (AUC) of GLPG3312 (μg.h/mL) (Part 4) | Between Day 1 pre-dose and Day 21
  To evaluate the pharmacokinetics (PK) of oral MAD of GLPG3312, in adult, healthy, subjects, when given as MR formulation
Terminal elimination half-life (t1/2) of GLPG3312 (h) (Part 1) | Between Day 1 pre-dose and Day 4
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3312, in adult, healthy, subjects, when given as IR formulation
Terminal elimination half-life (t1/2) of GLPG3312 (h) (Part 2) | Between Day 1 pre-dose and Day 7
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3312, in adult, healthy, subjects, when given as MR formulation
Terminal elimination half-life (t1/2) of GLPG3312 (h) (Part 4) | Between Day 1 pre-dose and Day 21
  To evaluate the pharmacokinetics (PK) of oral MAD of GLPG3312, in adult, healthy, subjects, when given as MR formulation
Cumulative amount of GLPG3312 excreted in urine (Aeurine)(mg) (Part 1) | Between Day 1 pre-dose and Day 4
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3312, in adult, healthy subjects, when given as IR formulation
Cumulative amount of GLPG3312 excreted in urine (Aeurine)(mg) (Part 2) | Between Day 1 pre-dose and Day 7
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3312, in adult, healthy, subjects, when given as MR formulation
Cumulative amount of GLPG3312 excreted in urine (Aeurine)(mg) (Part 4) | Between Day 1 pre-dose and Day 21
  To evaluate the PK of single and multiple ascending oral doses of GLPG3312, in adult, healthy subjects, when given as MR formulation.
Cumulative amount of GLPG3312 excreted in feces (Aefeces)(mg) (Part 4) | Between Day 1 pre-dose and Day 21
  To evaluate the PK of single and multiple ascending oral doses of GLPG3312, in adult, healthy subjects, when given as MR formulation.
Ratio in extent and exposure following dosing of GLPG3312 as MR formulation compared to following dosing as IR formulation, under fasted conditions (Part 1 versus Part 2) | Between Day 1 pre-dose and Day 4
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3312, in adult, healthy, subjects, when given as IR or as MR formulation
Ratio in extent and exposure following dosing of GLPG3312 as MR tablets under fed conditions (high-fat high calorie) versus fasted conditions (Part 3) | Between Day 1 pre-dose and Day 7
  To evaluate the food effect on the PK of a single oral dose of GLPG3312 in adult, healthy, subjects, when given as MR formulation

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Petkova, MD, Study Director — Galapagos NV
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

REFERENCES:
- [Derived] Temal-Laib T, Peixoto C, Desroy N, De Lemos E, Bonnaterre F, Bienvenu N, Picolet O, Sartori E, Bucher D, Lopez-Ramos M, Roca Magadan C, Laenen W, Flower T, Mollat P, Bugaud O, Touitou R, Pereira Fernandes A, Lavazais S, Monjardet A, Borgonovi M, Gosmini R, Brys R, Amantini D, De Vos S, Andrews M. Optimization of Selectivity and Pharmacokinetic Properties of Salt-Inducible Kinase Inhibitors that Led to the Discovery of Pan-SIK Inhibitor GLPG3312. J Med Chem. 2024 Jan 11;67(1):380-401. doi: 10.1021/acs.jmedchem.3c01428. Epub 2023 Dec 26. PMID 38147525